CLINICAL TRIAL: NCT04184349
Title: Truncal Ultrasound Guided Regional Anesthesia for Implantation and Revision of AICDs and Pacemakers in Pediatric Patients
Brief Title: Truncal Ultrasound Guided Regional Anesthesia for Implantation and Revision of Automatic Implantable Cardioverter Defibrillators (AICDs) and Pacemakers in Pediatric Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Olga Pawelek, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-19-0760
Record Dates: First submitted 2019-11-07; First posted 2019-12-03 (Actual); Results first posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Analgesia After Pacemaker; AICDS Implantation Pediatrics
Keywords: pacemaker; AICDS; regional anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Local Anesthetic (LA Group) (Active Comparator)
  Interventions: Drug: LA group
- B group (Active Comparator)
  Interventions: Drug: B Group

INTERVENTIONS:
Drug: LA group — In the LA group, only the local anesthetic infiltration will be performed by injecting the numbing medicine ropivacaine into the surgical site.
  Arms: Local Anesthetic (LA Group)
Drug: B Group — In the B Group,pectoral (PECS) and transversus thoracic plane(TTP) blocks will be performed by injecting the numbing medicine ropivacaine near the nerves.
  Arms: B group

SUMMARY:
The purpose of this study is to determine the efficacy and safety of truncal blocks for pacemaker and Automatic Implantable Cardioverter Defibrillator implantation in children and to prospectively evaluate whether there is a decrease in amount of narcotic medications need and track complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing implantation or revision of pacemaker or AICD in the pediatric cath lab

Exclusion Criteria:

* parent or patient refusal
* use of narcotic medications prior to procedure

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-06-09 (Actual); Study Completion 2022-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olga Pewelek, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Local Anesthetic (LA Group) | B Group
Started | 10 | 9
Completed | 10 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Local Anesthetic (LA Group) | B Group | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.10 (2.92) | 8.77 (3.96) | 11.05 (4.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 6
  Male | 9 | 4 | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: Total Narcotic Dose in Milligram Morphine Equivalents (MME) Per Kilogram
Time Frame: From 24 hours after procedure to 48 hours after procedure
Measure: Mean (Standard Deviation); unit: MME per kg
Arm/Group | Local Anesthetic (LA Group) | B Group
Number analyzed (Participants) | 10 | 9
MME per kg | 0.035 (0.082) | 0.008 (0.026)

2. Primary Outcome: Total Narcotic Dose in Milligram Morphine Equivalents (MME) Per Kilogram
Time Frame: up to 24 hours after procedure
Measure: Mean (Standard Deviation); unit: MME per kg
Arm/Group | Local Anesthetic (LA Group) | B Group
Number analyzed (Participants) | 10 | 9
MME per kg | 0.021 (0.044) | 0.008 (0.026)

3. Secondary Outcome: Pain as Measured by the Visual Analog Scale (VAS) Pain Score
Description: VAS pain scale is a range of scores from 0-100. A higher score indicates greater pain intensity.
Time Frame: up to 1.5 hours post procedure in post anesthesia care unit (PACU)
Population: Data were not collected for this outcome measure because this assessment was not used in the PACU. The Face, Legs, Activity, Cry, Consolability (FLACC) Pain Assessment Scale was used instead.
Arm/Group | Local Anesthetic (LA Group) | B Group
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Pain as Measured by the Visual Analog Scale (VAS) Pain Score
Description: VAS pain scale is a range of scores from 0-10. A higher score indicates greater pain intensity.
Time Frame: up to 24 hours post procedure
Population: Data were not collected from 1 participant in the Local Anesthetic (LA Group) arm because it was not charted by bedside nurse.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Local Anesthetic (LA Group) | B Group
Number analyzed (Participants) | 9 | 9
score on a scale | 1.33 (2.23) | 3.44 (3.46)

5. Secondary Outcome: Pain as Measured by the Face, Legs, Activity, Cry, Consolability (FLACC) Pain Assessment Scale
Description: Face, Legs, Activity, Cry, Consolability (FLACC) Pain Assessment measures pain with a total score that ranges from 0 to 10; a higher score indicating greater pain.
Time Frame: up to 6 hours post procedure in post anesthesia care unit (PACU)
Population: Data were not collected from 3 participants in the Local Anesthetic (LA Group) arm because it was not charted by bedside nurse. Data were not collected from 1 participant in the B group arm because it was not charted by bedside nurse.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Local Anesthetic (LA Group) | B Group
Number analyzed (Participants) | 7 | 8
score on a scale | 1.28 (2.36) | 1.62 (2.92)

6. Secondary Outcome: Number of Patients With the Incidence of Pruritis
Time Frame: up to 48 hours after procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Local Anesthetic (LA Group) | B Group
Number analyzed (Participants) | 10 | 9
Participants | 0 | 0

7. Secondary Outcome: Number of Patients With the Incidence of Nausea/Vomiting
Time Frame: up to 48 hours after procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Local Anesthetic (LA Group) | B Group
Number analyzed (Participants) | 10 | 9
Participants | 0 | 0

8. Secondary Outcome: Number of Patients With Respiratory Depression
Time Frame: up to 48 hours after procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Local Anesthetic (LA Group) | B Group
Number analyzed (Participants) | 10 | 9
Participants | 0 | 0

9. Secondary Outcome: Number of Patients With Local Anesthetic Toxicity
Time Frame: up to 48 hours after procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Local Anesthetic (LA Group) | B Group
Number analyzed (Participants) | 10 | 9
Participants | 0 | 0

10. Secondary Outcome: Number of Patients With Incidence of Pneumothorax
Time Frame: up to 48 hours after procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Local Anesthetic (LA Group) | B Group
Number analyzed (Participants) | 10 | 9
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 48 hours
Arm/Group | Local Anesthetic (LA Group) | B Group
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 0/10 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-19): https://cdn.clinicaltrials.gov/large-docs/49/NCT04184349/Prot_SAP_000.pdf